CLINICAL TRIAL: NCT04536051
Title: A Randomized, Controlled, Phase III Study to Determine the Safety, Efficacy, and Immunogenicity of the Non-Replicating ChAdOx1 nCoV-19 Vaccine
Brief Title: A Study of a Candidate COVID-19 Vaccine (COV003)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: COV003
Record Dates: First submitted 2020-09-01; First posted 2020-09-02 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-09

CONDITIONS: Coronavirus
Keywords: Covid-19; ChAdOx1 nCov19; sars-cov-2; vaccine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — ChAdOx1 nCoV-19; Acetaminophen; MenACWY

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1a: single dose ChAdOx & paracetamol (Experimental): Participants will receive a single standard dose of ChAdOx1 nCOV19 vaccine plus paracetamol
  Interventions: Biological: ChAdOx1 nCoV-19 single dose + paracetamol
- Group 1b: single dose MenACWY & paracetamol (Active Comparator): Participants will receive a single dose of MenACWY plus paracetamol
  Interventions: Biological: MenACWY single dose + paracetamol
- Group 1c: two dose ChAdOx & paracetamol (Experimental): Participants will receive two standard doses of ChAdOx1 nCoV-19 vaccine, 4-12 weeks apart, plus paracetamol
  Interventions: Biological: ChAdOx1 nCoV-19 two dose + paracetamol
- Group 1d: two dose MenACWy/saline & paracetamol (Active Comparator): Participants will receive MenACWY prime, and Saline Placebo boost (0.5mL) plus paracetamol
  Interventions: Biological: MenACWY prime & saline placebo boost + paracetamol

INTERVENTIONS:
Biological: ChAdOx1 nCoV-19 single dose + paracetamol — Single dose of ChAdOx1nCOV19 vaccine, 5x10^10 vp + paracetamol
  Arms: Group 1a: single dose ChAdOx & paracetamol
Biological: MenACWY single dose + paracetamol — Single dose of MenACWY + paracetamol
  Arms: Group 1b: single dose MenACWY & paracetamol
Biological: ChAdOx1 nCoV-19 two dose + paracetamol — Two dose of ChAdOx1 nCoV-19 vaccine, 5x10^10vp (prime) and 0.5mL boost (3.5 - 6.5 × 10^10 vp), 4-12 weeks apart + paracetamol
  Arms: Group 1c: two dose ChAdOx & paracetamol
Biological: MenACWY prime & saline placebo boost + paracetamol — MenACWY prime, and Saline Placebo boost (0.5mL) + paracetamol
  Arms: Group 1d: two dose MenACWy/saline & paracetamol

SUMMARY:
A Randomized, Controlled, Phase III Study to Determine the Safety, Efficacy, and Immunogenicity of the Non-Replicating ChAdOx1 nCoV-19 Vaccine.

DETAILED DESCRIPTION:
There will be 2 study groups and an anticipated enrolment of 10,300 health professionals and adults with high potential for exposure to SARS-CoV-2, aged ≥18 years.

All subjects will undergo follow-up for a total of 1 year post last vaccination. Additional visits or procedures may be performed at the discretion of the investigators, e.g., further medical history and physical examination, or additional blood tests and other investigations if clinically relevant

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 55 years of age
* Adults aged 56-69 years old (after review of safety data by DSMB in this age group in the UK trial)
* Adults aged 70 and above years old (after review of safety data by DSMB in this age group in the UK trial)
* Able and willing (in the Investigator's opinion) to fulfill all study requirements;
* Health professionals and adults at high risk of exposure to SARS-CoV-2, as defined in section 5.2 of this protocol;
* Serology with SARS-CoV-2 negative IgG antibodies; This inclusion criteria does not apply to participants enrolled from version 4.0 of the protocol onwards.
* Willing to allow investigators to discuss the participant's clinical history with their GP/personal physician and access medical records relevant to the study procedures
* Only for women of childbearing age willing to practice continuous effective birth control (see below) during the study, and a negative pregnancy test on the screening and vaccination day(s);
* Consent to abstain from blood donation during the course of the study;
* Provide informed consent in writing

Exclusion Criteria:

* Participation in trials of prophylactic drugs for COVID-19 during the course of the study; Note: Participation in COVID-19 treatment trials is permitted in case of hospitalization due to COVID-19, after confirmation of positive PCR. The study team should be informed as soon as possible. Participants with COVID-19 not hospitalized with positive PCR results for COVID-19 may be medicated according to standard clinical practice.
* Participation in SARS-CoV-2 serological research where participants are informed of their serological status during the course of the study;
* Planned receipt of any vaccine (authorized or investigational), within 30 days before and after vaccination;
* Prior receipt of an investigational vaccine or authorized with the possibility of impacting the interpretation of the study data (for example, vaccines vectorized by Adenovirus, any vaccines against coronavirus);
* Administration of immunoglobulins and/or any blood products in the three months prior to the planned administration of the candidate vaccine;
* Any confirmed or suspected immunosuppressive or immunodeficiency state; asplenia; severe recurrent infections and chronic use (more than 14 days) of immunosuppressive medication in the last 6 months, except for topical steroids or short-term oral steroids (cycle lasting ≤14 days);
* History of allergic disease or reactions possibly exacerbated by any component of ChAdOx1 nCoV-19 or MenACWY or paracetamol;
* Any history of angioedema;
* Any history of anaphylaxis;
* Pregnancy, lactation or willingness/intention to become pregnant during the study;
* Current diagnosis or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ);
* History of severe psychiatric illness that possibly affects your participation in the study;
* Hemorrhagic disorder (for example, factor deficiency, coagulopathy or platelet disorder), or a previous history of significant bleeding or bruising after IM injections or venipuncture;
* Current suspected or known dependence on alcohol or drugs;
* Severe and/or uncontrolled cardiovascular diseases, respiratory diseases, gastrointestinal diseases, liver disease, kidney disease, endocrine disorder, and neurological disease (mild/moderate well-controlled comorbidities are allowed);
* History of COVID-19 confirmed by laboratory;
* Seropositive for antibodies to SARS-CoV-2 before recruitment; This exclusion criteria does not apply to participants enrolled from version 4.0 of the protocol onwards
* Continued use of anticoagulants, such as coumarins and related anticoagulants (for example, warfarin) or new oral anticoagulants (for example, apixaban, rivaroxaban, dabigatran and edoxaban);
* Any other significant illness, disorder or finding that may significantly increase the risk for the participant, affect his/her ability to participate in the study or impair the interpretation of the study data.

Re-vaccination exclusion criteria (two-dose groups only)

* Anaphylactic reaction following administration of vaccine
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10300 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of ChAdOx1 nCoV-19 vaccine against COVID-19 disease confirmed with PCR | 12 months post final vaccination
  COVID-19 virologically confirmed symptomatic cases (PCR positive).

SECONDARY OUTCOMES:
Evaluate the safety, tolerability and reactogenicity profile of ChAdOx1 nCoV-19 candidate vaccine: occurrence of signs and symptoms of local and systemic reactogenicity requested during 7 days after vaccination | 7 days post vaccination
  Occurrence of signs and symptoms of local and systemic reactogenicity requested during 7 days after vaccination (in a subset of 200 participants)
Evaluate the safety, tolerability and reactogenicity profile of ChAdOx1 nCoV-19 candidate vaccine: occurrence of serious adverse events | 12 months post final vaccination
  Occurrence of serious adverse events
Evaluate the safety, tolerability and reactogenicity profile of ChAdOx1 nCoV-19 candidate vaccine: occurrence of episodes; intensified disease | 12 months post final vaccination
  Occurrence of episodes; intensified disease
Evaluate the efficacy of ChAdOx1 nCoV-19 candidate vaccine against severe and non-severe COVID-19 disease: hospitalization for COVID-19 disease confirmed by PCR | 12 months post final vaccination
  Hospitalization for COVID-19 disease confirmed by PCR
Evaluate the efficacy of ChAdOx1 nCoV-19 candidate vaccine against severe and non-severe COVID-19 disease: COVID-19 serious disease confirmed by PCR | 12 months post final vaccination
  COVID-19 serious disease confirmed by PCR
Evaluate the efficacy of ChAdOx1 nCoV-19 candidate vaccine against severe and non-severe COVID-19 disease: death associated with COVID-19 disease | 6 months
  Death associated with COVID-19 disease
Evaluate the efficacy of ChAdOx1 nCoV-19 candidate vaccine against severe and non-severe COVID-19 disease: antibodies against SARS-CoV-2 non-Spike protein (serum efficacy rates) | 12 months post final vaccination
  Antibodies against SARS-CoV-2 non-Spike protein (serum efficacy rates).
Evaluate the humoral immunogenicity of ChAdOx1 nCoV-19: antibodies against the SARS-CoV-2 spike protein (serum conversion rates) | 12 months post final vaccination
  Antibodies against the SARS-CoV-2 spike protein (serum conversion rates)
Evaluate the humoral immunogenicity of ChAdOx1 nCoV-19: virus neutralizing antibodies (NAb) against live and/or pseudotyped SARS-CoV-2 virus | 12 months post final vaccination
  Virus neutralizing antibodies (NAb) against live and/or pseudotyped SARS-CoV-2 virus
Assess the cellular immunogenicity of ChAdOx1 nCoV-19 candidate vaccine | 12 months post final vaccination
  Interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, Prof, Principal Investigator — University of Oxford
Locations (6):
- Brazil (6):
  - Instituto D'Or de Pesquisa e Ensino - I'Dor, Salvador, Estado de Bahia
  - Centro de Pesquisas Clinicas de Natal (CPCLIN), Natal, Rio Grande do Norte
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Santa Maria (UFSM), Santa Maria, Rio Grande do Sul
  - Instituto D'Or de Pesquisa e Ensino - I'Dor, Rio de Janeiro
  - CRIE, Universidade Federal de São Paulo, São Paulo

REFERENCES:
- [Derived] Costa Clemens SA, Bibi S, Marchevsky NG, Aley PK, Cappuccini F, Davies SA, Gonzalez I, Kelly SC, Mujadidi YF, Pipolo Milan E, Schwarzbold AV, Sprinz E, Voysey M, Weckx LY, Wright D, Bansal H, Bergagard MAS, Isaacs AJ, Kelly EJ, Lan D, Morgan S, Shankar NK, Shoemaker K, Villafana TL, Lambe T, Green JA, Pollard AJ. Immunogenicity and Safety of ChAdOx1 nCoV-19 (AZD1222) as a Homologous Fourth-Dose Booster: A Substudy of the Phase 3 COV003 Trial in Brazil. Mayo Clin Proc Innov Qual Outcomes. 2025 Jul 11;9(4):100642. doi: 10.1016/j.mayocpiqo.2025.100642. eCollection 2025 Aug. PMID 40686533
- [Derived] Conlin K, Jenkin D, de Whalley P, Weckx LY, Folegatti PM, Bibi S, Lambe T, Aley PK, Pollard AJ, Voysey M, Costa Clemens SA; COV003 Study Group. Predictors of severity of SARS-CoV-2 infections in Brazil: Post hoc analyses of a randomised controlled trial. Vaccine. 2025 Jan 25;45:126582. doi: 10.1016/j.vaccine.2024.126582. Epub 2024 Dec 14. PMID 39675209